CLINICAL TRIAL: NCT03405103
Title: Efficacy of m-Health Self-Management Intervention
Brief Title: Striving to be Strong: Self-management
Acronym: S2BS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: Marquette University (Other); Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Polly Ryan, PhD, RN, FAAN, Researcher, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01NR013913-01 (NIH)
Record Dates: First submitted 2018-01-06; First posted 2018-01-19 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Osteoporosis; Health Behavior
Keywords: self-management; m-Health
MeSH Terms: conditions — Osteoporosis; Health Behavior

STUDY DESIGN:
Intervention Model Description: Repeated measures randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Striving (Experimental): Striving vs Boning-up & Personal Choice
  Interventions: Behavioral: Striving
- Boning-up Standard Education (Active Comparator): Boning-up vs Striving and Personal Choice
  Interventions: Behavioral: Boning-Up
- Personal Choice (Sham Comparator): Personal Choice vs Striving & Boning-up
  Interventions: Behavioral: Personal Choice

INTERVENTIONS:
Behavioral: Striving
  Other Names: S2BS
  Arms: Striving
Behavioral: Boning-Up
  Arms: Boning-up Standard Education
Behavioral: Personal Choice
  Arms: Personal Choice

SUMMARY:
The vast majority of people want to be healthy and often make a change to be healthier. Change that is begun is seldom maintained. Osteoporosis is an example of one condition where people are encouraged to regularly engage in preventative health behaviors. This is a study testing a new approach to helping women engage in osteoporosis health behaviors. This new approach includes beliefs, self-regulating skills and abilities, and social facilitation delivered via a cell phone app. If effective, this approach could be tested with other health behaviors.

DETAILED DESCRIPTION:
The goal of this project is to test the efficacy a theory based, patient-centered, dynamically tailored intervention delivered via a cell phone app. The four aims of this project are to: 1) Test the efficacy of the intervention to improve long term maintenance of osteoporosis prevention health behaviors in midlife women, 2) evaluate moderators and mediators of long-term engagement in health behaviors, 3) describe processes of health behavior change and evaluate differences within and between subjects using Ecological Momentary Assessments (EMA) as a complement to traditional measures and 4) evaluate the utility of The Individual and Family Self-Management Theory to explain health behavior change. In the U.S., over 35 million women either have or are at high risk for osteoporosis at an anticipated cost of greater than $25 billion by 2025. Osteoporosis affects 1 out of 2 White women, is rapidly growing among populations of color and causes high chronic disease burden worldwide. Less than 6% of women regularly engage in the basic health promotion behaviors. The vast disparity between the high prevalence of osteoporosis and the low number of people who engage in preventative care highlights this condition as one of many striking examples of the crucial role behavior change could play in improving health and decreasing health care costs. New knowledge suggests enhancing knowledge and beliefs, self-regulation skill and abilities, and social facilitation leads to self-management and improved health outcomes. It is hypothesized that the more an intervention integrates health behavior change processes into daily activities the more likely it is to increases one's capacity to self-manage. The work proposed is significant because it focuses on the serious and prevalent condition of osteoporosis; tests the application of a theory based, patient-centered, dynamic intervention designed to improve outcomes; and, decisively bundles new knowledge about methodologies, intervention processes, and delivery media to provide a cohesive foundation for intervention development and testing. Innovative aspects include use of EMAs as a complementary approach to providing feedback and measuring behavior change processes; testing a newly identified health behavior change theory; and development and evaluation of a cell phone app, one type of m-Health. Through technological advances we now have the capacity to integrate health behavior change processes into every day activities via a cell phone app but the effectiveness of the app to change health behaviors has not been demonstrated empirically. A three-group randomized controlled longitudinal design with data collected at baseline, 3, 6, 9, and 12 months will be used. A convenience sample of 288 (96 per group) community dwelling women will be enrolled. Outcomes will be evaluated with self-report, behavioral performance, and bio-behavioral measures, including DXA and vitamin D. The expected outcomes are achievement of an increase in women's initiation and long term maintenance of osteoporosis self-management behaviors and stabilization of bone mineral density.

ELIGIBILITY:
Inclusion Criteria:

* healthy (able to participate in physical activity, not receiving medical care for chronic condition, not taking medications that would affect bone, greater than 5 years post treatment for cancer) not pregnant or lactating speaks and reads English consumes at least 200 mg less recommended amount of dietary calcium

Exclusion Criteria:

* diagnosis of osteoporosis, history of fragile fracture, does not engage in vigorous activity more than 2 times a week

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 290 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mineral Density | Baseline and 12 months
  Bone Mineral Density obtained via Dual Energy x-ray absorptiometry

SECONDARY OUTCOMES:
Calcium Focused Food Diary | Baseline, 3, 6, 9, and 12 months
  mg of calcium obtained via food as measured by Calcium Focused Food Diary. Calculated daily for 3-days. Total mg of calcium across 3 measurement days used .
Physical Activity Questionnaire (IPAQ)- Short Form: Measure of time and intensity of persons engagement in physical activity. | Baseline, 3, 6, 9, and 12 months
  Self-report of frequency and intensity of engagement in common leisure time (non-work related) Physical Activites. Calculated score accounts for time and METs. Data are collected over a 7-day period of time across pre-specified categories of leisure time activities and total score calculated by adding totals obtained for each day. Sub-totals of low, medium, and vigorous activities. Higher the score is associated with higher level of activities.
Balance | Baseline and 12 months
  4 stage Balance Test: Ability to hold one of four positions for 45 seconds. Positions inclue eyes open, both feet on ground: eyes closed both feet on ground: eyes open, one foot on ground; eyes closed, one foot on ground. Scored by adding total seconds across 4 positions.
Stand Test | Baseline and 12 months
  Leg strength: time it takes participant to stand and sit ten times, Measured in seconds.
6-minute walk test | Baseline and 12 months
  Functional Status: measure of distance walked in 6 minutes. Measured in feet and inches
Functional Movement Screen (adaptation) | Baseline and 12 months
  Strength and Balance. Test includes four movements specifically hurdle step, in-line lunge, straight leg raise, and squat. All movements were video taped from two positions (front and side). Certified professionals evaluated the videoed four movement and scored each movement using a standardized scoring template. Individual scores are obtained for each of the four movement and a total score is obtained by adding the scores from the four movements. Scores for each movement include 0=pain and score of 1-3 with 3 indicating the best performance.
Engagement in Self-regulation processes: "What are you doing today"/ DOTs | Over 12 months a total of 284 text message were sent to each participant via newly designed app. Score included frequency of behavior and self-regulation process for 4 week periods over 12 months.
  Ecological Momentary Assessments. Osteoporosis prevention focuses on four behaviors: calcium intake, balance, core and leg strength, and physical activity. For each of the four behaviors the participant indicates (using a yes or no response) if they engaged in any of the self-regulation processes (e.g., setting a goal, making a plan, engaging in the behavior, monitoring) for each of the 4 behaviors (calcium, balance, strength, and physical activity.
  For each of these four behaviors participants select all of the component of the Self-regulation process
vitamin D | Baseline and 12 months
  serum vitamin D level measured in nmole/L

CONTACTS AND LOCATIONS:
Overall Officials: Polly A Ryan, PhD, Principal Investigator — University of Wisconsin, Milwaukee

IPD SHARING:
Plan to Share IPD: Undecided
Undecided